CLINICAL TRIAL: NCT03709784
Title: A Prospective, Multi-center, Observational Study of the Safety, Tolerability and Effectiveness of SPINRAZA® (Nusinersen) in Adult Patients With Spinal Muscular Atrophy
Brief Title: Spinraza in Adult Spinal Muscular Atrophy
Acronym: SAS
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201805187
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Spinal Muscular Atrophy; Spinal Muscular Atrophy Type II; Spinal Muscular Atrophy Type 3
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5cc of Cerebral Spinal Fluid (CSF) is collected and typically discarded as part of the typical clinical encounter when SPINRAZA® (nusinersen) is administered. This 5cc of CSF will be collected for research purposes at each dosing visit. Blood samples, including whole blood, serum, and plasma (3 teaspoons total) will be collected within seven days of standard of care SPINRAZA® (nusinersen) administration at dose #1, 2, 4, 5, 7, 9 and 11.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cohort 1: This is a prospective, longitudinal, multi-center, observational study designed to evaluate the safety, tolerability, and effectiveness of SPINRAZA® (nusinersen) in ambulatory and non-ambulatory adult patients with SMA. Subjects with SMA II/III that are 18 years to 70 years of age who are planning to initiate treatment with SPINRAZA® (nusinersen) as part of their clinical care plan will be enrolled in this study. This study does not provide SPINRAZA® (nusinersen) or cover costs associated with standard clinical care.These patients will be treated by their respective physicians according to standard clinical practice. Study visits, some of which including standardized assessments of strength and function, will occur at baseline, day 15 after treatment initiation, day 30, day 60, and then 4-month intervals through month 30.
  Interventions: Drug: Observational study to examine safety, tolerability, and effectiveness of SPINRAZA® prescribed as part of standard of care
- Cohort 2: The cohort 2 is a one time survey to gain a better understanding of this adult population and their treatment preferences.
  Interventions: Other: One time survey

INTERVENTIONS:
Drug: Observational study to examine safety, tolerability, and effectiveness of SPINRAZA® prescribed as part of standard of care — This is an observational study of adult patients with SMA to examine the safety, tolerability, and effectiveness of SPINRAZA® (nusinersen) for up to 30 months.
  Groups: Cohort 1
Other: One time survey — One time survey
  Groups: Cohort 2

SUMMARY:
This is a longitudinal, observational study of adult patients with genetically confirmed chromosome 5q SMA to examine the safety, tolerability, and effectiveness of SPINRAZA® (nusinersen) for up to 30 months.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, multi-center, observational study designed to evaluate the safety, tolerability, and effectiveness of SPINRAZA® (nusinersen) in ambulatory and non-ambulatory adult patients with SMA. Subjects with SMA II/III that are 18 years to 70 years of age who are planning to initiate treatment with SPINRAZA® (nusinersen) as part of their clinical care plan will be enrolled in this study. This study does not provide SPINRAZA® (nusinersen) or cover costs associated with standard clinical care.These patients will be treated by their respective physicians according to standard clinical practice. Study visits, some of which including standardized assessments of strength and function, will occur at baseline, day 15 after treatment initiation, day 30, day 60, and then 4-month intervals through month 30.

After 30 months an additional cohort 2 was added. The approval date was March 13, 2023. The cohort 2 is a one time survey to gain a better understanding of this adult population and their treatment preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Males and females with SMA type II or type III, aged 18 to 70 years at the time of enrollment.
3. Genetic documentation of 5Q SMA homozygous gene deletion, mutation, or compound heterozygote.
4. Are treatment naïve for SPINRAZA® (nusinersen).
5. Have been prescribed SPINRAZA® (nusinersen) by the treating physician as part of their clinical care for SMA following the FDA approved prescribing information guidelines as follows: dose level (12 mg), dosing schedule (3 loading doses administered at 14-day intervals, and the fourth loading dose administered 30 days after the third dose and subsequent maintenance doses administered every 4 months) and safety lab monitoring (CBC, PT, INR, PTT, UA) done prior to each dose administration.
6. Believed to be able to complete all study procedures, measurements and visits.
7. Estimated life expectancy at least 30 months from first dosing, in the opinion of the Investigator.
8. Revised upper limb module (RULM) score ≥ 4 (more than marginal upper extremity function/strength.
9. Must meet either Group 1 or Group 2 criteria.

For Group 1 subjects:

1. May be ambulatory or non-ambulatory (defined as being wheelchair reliant at least 75% of time and unable to walk at least 10 meters without assistance).
2. RULM score of 4-34, inclusive.

For Group 2 subjects:

1. Ability to walk at least 10 meters without assistance (i.e., four point walking aid).
2. Be free of major orthopedic deformities that limit ambulation.
3. An ambulatory subject can qualify for both Group 1 and Group 2 if the RULM score is ≤ 34.

Exclusion Criteria:

1. Revised upper limb score ≤ 3.
2. Respiratory insufficiency, defined by the medical necessity for invasive or noninvasive ventilation for >16 hours during a 24-hour period, at screening.
3. Hospitalization for major medical event including: surgery (i.e., scoliosis surgery, other surgery), cardiac event, pulmonary event, or other major medical problem within 2 months of screening or planned major surgical procedure likely to impact the clinical assessments during the duration of the study. Outpatient surgical procedure (i.e., placement of feeding tube) is not considered an exclusionary major medical event.
4. Presence of a symptomatic severe active infection or illness during the screening period that is likely to impact the performance on the clinical assessments.
5. Prior exposure to SPINRAZA® (nusinersen).
6. Prior disorder, injury (e.g., upper or lower limb fracture) or surgical procedure which impacts the subject's ability to perform any of the outcome measure testing required in the protocol and from which the subject has not fully recovered or achieved a stable baseline.
7. Treatment with an investigational drug (e.g., oral albuterol/salbutamol, riluzole, carnitine, creatine, sodium phenylbutyrate, etc.), biological agent, or device within 1-month of Screening or 5 half-lives of study agent, whichever is longer. Patients using intrathecal drug delivery devices, including investigational devices with an active IDE designation in the United States, may be eligible but require Study PI approval prior to enrollment.
8. Any history of exposure to gene therapy, antisense oligonucleotide therapy, or cell transplantation that was intended for the treatment of SMA.
9. Ongoing medical condition that according to the Clinical Center Investigator would interfere with the conduct and assessments of the study. Examples are medical disability (e.g., wasting or cachexia, severe anemia, etc.) that would interfere with the assessment of safety or would compromise the ability of the subject to undergo study procedures.

For Cohort 2 Inclusion criteria

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Males and females with SMA type II or type III, aged 18 to 70 years at the time of enrollment.
3. Genetic documentation of 5Q SMA homozygous gene deletion, mutation, or compound heterozygote.
4. Believed to be able to complete the structured interview.

Cohort 2 Exclusion Criteria

1. Ongoing medical condition that according to the Clinical Center Investigator would interfere with the conduct and assessments of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with SMA that are 18 years to 70 years of age who are planning to initiate treatment with SPINRAZA® (nusinersen) as part of their clinical care plan.
  For Cohort 2 - Subjects with SMA that are 18 years to 70 years with SMA type II/III.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the 6-Minute Walk Test (6MWT) for ambulatory SMA patients | 30 months
  Assess effectiveness of SPINRAZA® (nusinersen) treatment on mobility and ambulation in ambulatory adult SMA patients, comparing changes in total distance walked in in six minutes from baseline until end of treatment at 30 months..
Change from baseline in Revised Upper Limb Module (RULM) for weak ambulatory and non-ambulatory SMA patients | 30 months
  Assess the effectiveness of SPINRAZA® (nusinersen) treatment on upper extremity function in ambulatory and non-ambulatory adult SMA patients, comparing change in RULM score from baseline until end of treatment at 30 months.

SECONDARY OUTCOMES:
To describe the demographic and clinical characteristics, disease burden, treatment preferences, and subjective assessments of disease progression | 6 months to 1 year
  One time survey

CONTACTS AND LOCATIONS:
Overall Officials: Craig Zaidman, MD, Principal Investigator — Washington University School of Medicine
Locations (11):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital-Harvard University, Boston, Massachusetts
  - Memorial Healthcare, Owosso, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Houston Methodist Neurological Institute, Houston, Texas
  - Children's Hospital of the King's Daughthers, Norfolk, Virginia
  - University of Washington, Seattle, Washington
- Montreal Neurological Institute and Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Vivo DC, Bertini E, Swoboda KJ, Hwu WL, Crawford TO, Finkel RS, Kirschner J, Kuntz NL, Parsons JA, Ryan MM, Butterfield RJ, Topaloglu H, Ben-Omran T, Sansone VA, Jong YJ, Shu F, Staropoli JF, Kerr D, Sandrock AW, Stebbins C, Petrillo M, Braley G, Johnson K, Foster R, Gheuens S, Bhan I, Reyna SP, Fradette S, Farwell W; NURTURE Study Group. Nusinersen initiated in infants during the presymptomatic stage of spinal muscular atrophy: Interim efficacy and safety results from the Phase 2 NURTURE study. Neuromuscul Disord. 2019 Nov;29(11):842-856. doi: 10.1016/j.nmd.2019.09.007. Epub 2019 Sep 12. PMID 31704158
- [Background] Finkel RS, Mercuri E, Darras BT, Connolly AM, Kuntz NL, Kirschner J, Chiriboga CA, Saito K, Servais L, Tizzano E, Topaloglu H, Tulinius M, Montes J, Glanzman AM, Bishop K, Zhong ZJ, Gheuens S, Bennett CF, Schneider E, Farwell W, De Vivo DC; ENDEAR Study Group. Nusinersen versus Sham Control in Infantile-Onset Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1723-1732. doi: 10.1056/NEJMoa1702752. PMID 29091570
- [Background] Mercuri E, Darras BT, Chiriboga CA, Day JW, Campbell C, Connolly AM, Iannaccone ST, Kirschner J, Kuntz NL, Saito K, Shieh PB, Tulinius M, Mazzone ES, Montes J, Bishop KM, Yang Q, Foster R, Gheuens S, Bennett CF, Farwell W, Schneider E, De Vivo DC, Finkel RS; CHERISH Study Group. Nusinersen versus Sham Control in Later-Onset Spinal Muscular Atrophy. N Engl J Med. 2018 Feb 15;378(7):625-635. doi: 10.1056/NEJMoa1710504. PMID 29443664